CLINICAL TRIAL: NCT06632743
Title: Sarcopenia in Cirrhosis and Chronic Inflammatory Bowel Disease: An Austrian Biobanking Study
Brief Title: Austrian Biobanking Study for Sarcopenia
Acronym: ASGSC
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 34-294 ex 21/22
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Sarcopenia
Keywords: Register; Biosamples; Microbiome
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Plasma, Serum, Stool, Urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sarcopenia: Diagnosed with sarcopenia according to EWGSOP (European Working Group on Sarcopenia in Older People)
- no sarcopenia: Not fulfilling sarcopenia criteria according to EWGSOP

SUMMARY:
The investigators aim to set up a biobanking study in Graz, Austria, to study sarcopenia in liver cirrhosis and chronic inflammatory bowel disease by collecting a standardized dataset including routine clinical and biochemical tests; biosamples to assess novel biomarker as well as advanced clinical assessments. In a small country like Austria, a nationwide biobanking study can enhance research enormously. The investigators therefore aim to extend the registry to all tertiary liver care centers in Austria in a second step.

DETAILED DESCRIPTION:
As the average age of societies rises, so too does the onset of debilitating diseases. Among these, sarcopenia, which is defined as a progressive decline in muscle mass, quality and strength, affects over one third and of people above 70 and half of patients with chronic diseases- such as liver cirrhosis or chronic inflammatory bowel disease (IBD). Sarcopenia remains an unmet clinical need with wide reaching implications affecting patients, their families and the health care system as a whole whereby patients lose independence due to their frailty which consequently decreases overall life quality and increases the risk of severe injuries, and complication thereof, due to falls.The pathogenesis of sarcopenia in cirrhosis is incompletely understood: Decreased protein synthesis and increased protein degradation mediated by inflammation contribute to sarcopenia in cirrhosis. In chronic inflammatory bowel disease, sarcopenia often results from a complex interplay of various factors, including inflammation, malabsorption, limited physical activity, and nutrient deficiencies.

Despite the high prevalence of sarcopenia among the aging and diseased populations, its diagnosis remains challenging as generally accepted international standards are lacking. Combined with the low agreement of available diagnosis criteria, this further complicates diagnostic methods. (8) To date, the diagnosis of sarcopenia relies on the quantification of muscle mass and a clinical assessment of muscle strength. For the estimation of muscle mass, costly computed tomography (CT) or magnetic resonance imaging (MRI) are the methods of choice to quantify the muscled area of a cross section on the level of the L3 vertebra- these methods also require skilled personnel and specialized software solutions for image evaluation. Methods used to assess muscle function, such as hand grip strength, gait speed and knee flexion/extension also require skilled personnel and present an additional layer of complexity to the overall diagnosis as they are difficult to standardize and heavily dependent patient compliance. Furthermore, the interpretation of the outlined diagnostic measures remains ambiguous, since different consensus definitions show conflicting results in different patient populations. Biomarker of muscle function and inflammation, as well as hormone assessments have been considered as useful diagnostic alternatives, however they are not part of clinical routine yet. Taken together, current diagnostic options for sarcopenia remain grossly insufficient which, often, allows this detrimental condition to be missed in clinical practice thereby hindering adequate and timely intervention.

In addition, currently there is no medical treatment available for sarcopenia. The current recommendation therefore is to improve nutrition, especially regarding the protein content, and physical activity.

Acquiring large enough datasets is of utmost importance to validate diagnostic tools or develop novel biomarker and therapies.

ELIGIBILITY:
Inclusion Criteria:

* Age >18y
* Informed consent
* CT/MRI scan as part of routine care within +/-2 month of the study visit

Exclusion Criteria:

* Hepatic encephalopathy > grade 2 and or other cognitive disorder not allowing informed consent
* Hepatocellular carcinoma stage BCLC C or D
* Any other condition or circumstance, which, in the opinion of the investigator, would affect the patient's ability to participate in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical/radiological/histological diagnosis of cirrhosis or chronic liver disease or histological diagnose of chronic inflammatory bowel disease
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2033-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Austrian-wide sarcopenia register | At enrolment
  Recruitment of 1000 people with/without sarcopenia

OTHER OUTCOMES:
Diagnostic accuracy | At enrolment
  Comparison of diagnostic accuracy of different published methods for sarcopenia diagnosis
Cut off definition | At enrolment
  Development of cut offs for well-established and novel biomarker for sarcopenia
AI (artificial intelligence) guided sarcopenia diagnosis | At enrolment
  Training of a neuronal network to distinguish between face pictures of patients with and without sarcopenia
Hypothesis generation | At enrolment
  Development of hypotheses for new diagnostic tools and interventional studies

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available in a public repository after the study is completed
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1.1.2035 unlimited